CLINICAL TRIAL: NCT06572111
Title: A Phase I, Open-label Trial to Investigate the Metabolism, Pharmacokinetics (Following a Mass Balance Design; Part A) and Absolute Bioavailability of BI 1839100 (C-14) After Oral and Intravenous Administration (Part B) in Healthy Male Subjects
Brief Title: A Study in Healthy Men to Test How BI 1839100 is Taken up and Handled by the Body
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Company decision
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1490-0006; 2024-510870-26-00 (Registry Identifier: CTIS); U1111-1308-5227 (Other: WHO International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2024-08-23; First posted 2024-08-26 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Healthy
MeSH Terms: interventions — Carbon-14

STUDY DESIGN:
Intervention Model Description: Part A: open-label, single arm, single-dose Part B: non-randomized, open-label, single-arm, single period, fixed sequence, crossover
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part A: BI 1839100 (C-14) formulation 1 (Experimental): BI 1839100 (C-14) = BI 1839100 Carbon 14 Radiolabelled
  Interventions: Drug: BI 1839100 (C-14) formulation 1
- Part B: BI 1839100 followed by BI 1839100 (C-14) formulation 2 (Experimental)
  Interventions: Drug: BI 1839100; Drug: BI 1839100 (C-14) formulation 2

INTERVENTIONS:
Drug: BI 1839100 (C-14) formulation 1 — BI 1839100 (C-14) formulation 1
  Arms: Part A: BI 1839100 (C-14) formulation 1
Drug: BI 1839100 — BI 1839100
  Arms: Part B: BI 1839100 followed by BI 1839100 (C-14) formulation 2
Drug: BI 1839100 (C-14) formulation 2 — BI 1839100 (C-14) formulation 2
  Arms: Part B: BI 1839100 followed by BI 1839100 (C-14) formulation 2

SUMMARY:
This trial is conducted in healthy male subjects to evaluate the drug BI 1839100. The trial has two main parts. Part A aims to understand how BI 1839100 is processed in the body after an oral dose. It measures the total recovery of the drug and its radioactive label in urine and feces. It also determines the concentrations in blood plasma and investigates the drug's metabolic pathways. Part B aims to compare the absolute bioavailability of BI 1839100 when administered orally and intravenously.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electronic cardiogram (ECG), and clinical laboratory tests.
2. Age of 18 to 59 years (inclusive at screening)
3. Body mass index (BMI) of 18.5 to 30.0 kg/m2 (inclusive at screening)
4. Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial

Exclusion Criteria:

1. Any finding in the medical examination (including blood pressure (BP), pulse rate (PR), or ECG that deviates from normal and is assessed as clinically significant by the investigator
2. Repeated measurement of systolic BP outside the range of 90 to 140 mmHg, diastolic BP outside the range of 50 to 90 mmHg, or PR outside the range of 45 to 90 bpm (subjects with PR values between 45 and 50 bpm may only be enrolled in case they have normal thyroid function (thyroid-stimulating hormone (TSH) and free thyroxine (FT4) at baseline-screening, no clinical symptoms associated with the bradycardia and no apparent signs of other diseases causing bradycardia such as hypothyroidism or heart conduction abnormalities)
3. Any laboratory value outside the reference range that the investigator considers to be of clinical significance
4. Any evidence of a concomitant disease assessed as clinically significant by the investigator
5. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders assessed as clinically significant by the investigator
6. Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the Pharmacokinetics (PKs) of the trial medication (except appendectomy or simple hernia repair)
7. Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders assessed as clinically relevant by the investigator
8. History of significant orthostatic hypotension, fainting spells, or blackouts Further exclusion criteria apply.

Ages: 18 Years to 59 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2024-09-30 (Actual); Primary Completion 2024-10-28 (Actual); Study Completion 2025-09-02 (Actual)

PRIMARY OUTCOMES:
Mass balance and total recovery of [C-14]-radioactivity in urine and feces. | From drug administration up to Day 21.
  Part A
Area under the concentration-time curve of Carbon-14-labeled BI 1839100 after intravenous administration and BI 1839100 after oral administration, extrapolated to infinity (AUC0-∞). | From drug administration up to Day 21.
  Part B

SECONDARY OUTCOMES:
Maximum measured concentration of BI 1839100 and Carbon-14-labeled BI 1839100 in plasma (Cmax). | Two hours before drug administration up to Day 21.
  Part A
Area under the concentration-time curve of BI 1839100 and Carbon-14-labeled BI 1839100 from 0 to the last quantifiable time point (AUC0-tz). | Two hours before drug administration up to Day 21.
  Part A
Area under the concentration-time curve of Carbon-14-labeled BI 1839100 in plasma after intravenous administration and BI 1839100 after oral administration, from 0 to the last quantifiable time point (AUC0-tz). | Two hours before drug administration up to 72 hours (Day 4).
  Part B
Maximum measured concentration of Carbon-14-labeled BI 1839100 in plasma after intravenous administration and BI 1839100 after oral administration (Cmax). | Two hours before drug administration up to 72 hours (Day 4).
  Part B

CONTACTS AND LOCATIONS:
Locations (1):
- ICON-Groningen-62040, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com